CLINICAL TRIAL: NCT04774718
Title: A Phase I/II, Open-Label, Multicenter, Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Alectinib in Pediatric Participants With ALK Fusion-Positive Solid or CNS Tumors for Whom Prior Treatment Has Proven to be Ineffective or for Whom There is No Satisfactory Treatment Available
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Alectinib in Pediatric Participants With ALK Fusion-Positive Solid or CNS Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO42286; 2020-004239-25 (EudraCT Number)
Record Dates: First submitted 2021-02-10; First posted 2021-03-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ALK Fusion-positive Solid or CNS Tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALK-Fusion Positive (Experimental): Part 1 is a dose-confirmation phase to confirm the recommended phase 2 dose (RP2D). In Parts 2 and 3, participants will receive alectinib at the RP2D on Days 1-28 of each 28-day cycle
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive twice-daily alectinib capsules on Days 1-28 of each 28-day cycle

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and efficacy of alectinib in children and adolescents with ALK fusion-positive solid or CNS tumors for whom prior treatment has proven to be ineffective or for whom there is no satisfactory standard treatment available.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed diagnosis of CNS or solid tumors with documented evidence of ALK gene fusions as assessed centrally through the use of the investigational F1CDx assay or based on pre-existing NGS test results
* Disease status: prior treatment proven to be ineffective (i.e. relapsed or refractory), or for whom there is no satisfactory standard treatment available. Disease should be measurable and evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1, or Response Assessment in Neuro-oncology criteria (RANO) +/- bone marrow criteria for primary CNS tumors or International Neuroblastoma Response Criteria (INRC)
* Available tumor tissue for submission to the Sponsor from active disease, obtained subsequent to last anti-cancer therapy regimen administered and obtained prior to study enrollment (preferred option), or archival tumor tissue from original diagnosis, or willingness to undergo a core or excisional biopsy sample collection prior to enrollment
* For participants < 16 years old, Lansky Performance Status >/= 50%
* For participants >/= 16 years old, Karnofsky Performance Status >/= 50%
* Adequate bone marrow function as defined by the protocol within at least 28 days prior to initiation of study drug
* Participant and/or caregiver willingness and ability to complete clinical outcome assessments throughout the study using either electronic, paper, or interviewer methods
* For females of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs, as defined by the protocol
* For males who are not surgically sterile: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating sperm, as defined by the protocol

Exclusion Criteria

* Medical history of: prior use of ALK inhibitors; diagnosis of Anaplastic Large Cell Lymphoma (ALCL); any gastrointestinal disorder that may affect absorption of oral medications, such as mal-absorption syndrome or status post-major bowel resection; history of organ transplant; stem cell infusions as defined by the protocol
* Substance abuse within 12 months prior to screening
* Familial or personal history of congenital bone disorders, bone metabolism alterations, or osteopenia
* Treatment with investigational therapy 28 days prior to initiation of study drug
* Liver or kidney disease as defined by the protocol
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade >/=3 toxicities attributed to any prior therapy such as radiotherapy (excluding alopecia), which have not shown improvement and are strictly considered to interfere with alectinib
* Co-administration of anti-cancer therapies other than those administered in this study
* Active hepatitis B or C virus (HBV, HBC), or known HIV-positivity or AIDS-related illness
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the Principal Investigator, pose an unacceptable risk to the participant in this study
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; such conditions should be discussed with the participant before trial entry
* Planned procedure or surgery during the study except as permitted treatment as defined by the protocol
* Infection considered by the investigator to be clinically uncontrolled or of unacceptable risk to the participant upon induction of neutropenia, including participants who are, or should be, on antimicrobial agents for the treatment as active infection
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of alectinib

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2032-02-28 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Participants with Dose-Limited Toxicities (DLTs) | Cycle 1 (cycle length = 28 days)
Percentage of Participants with Adverse Events | Up to 10 years
Plasma Concentration of Alectinib | Up to 10 years
Plasma Concentration of Alectinib Metabolite (M4) | Up to 10 years
Confirmed Objective Response Rate (ORR): Defined as the Proportion of Participants with Complete Response (CR) or Partial Response (PR) on two Consecutive Occasions >/= 4 Weeks Apart, as Determined by Blinded Independent Central Review (BICR) | Up to 10 years

SECONDARY OUTCOMES:
Confirmed ORR as Determined by the Investigator | Up to 10 years
Duration of Response (DOR) as Determined by BICR and the Investigator | From the first occurrence of a documented objective response (CR or PR) to disease progression or death from any cause, whichever occurs first (up to 10 years)
Time to Response (TTR) as Determined by BICR and the Investigator | From the first dose of alectinib to the first documentation of objective response (CR or PR) (up to 10 years)
Clinical Benefit Rate (CBR) as Determined by BICR and the Investigator | 6 months after the first dose of alectinib
Progression-Free Survival (PFS) as Determined by BICR and the Investigator | From the first dose of alectinib to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 10 years)
Overall Survival (OS) | From the first dose of alectinib to the date of death due to any cause (up to 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (33):
- United States (7):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Jude Children'S Research Hospital, Memphis, Tennessee
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
- Brazil (2):
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Graacc-Grupo de Apoio ao adolescente e a crianca com cancer, São Paulo, São Paulo
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- China (2):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
- Rigshospitalet, København Ø, Denmark
- France (3):
  - Centre Léon Bérard, Institut d?Hémato-Oncologie Pédiatrique, Lyon
  - Hôpital de la Timone, Oncologie Pédiatrique, Marseille
  - Institut Curie - Centre de Lutte Contre le Cancer (CLCC) de Paris, Paris
- Universitätsklinikum Heidelberg, Heidelberg, Germany
- Italy (3):
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS, Genoa, Liguria
  - Istituto Nazionale Tumori di Milano, Milan, Lombardy
  - Dipartimento di Scienze Pediatriche Adolescenza, Turin, Piedmont
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - Great Ormond Street Hospital, London
  - Royal Manchester Childrens Hospital, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing